CLINICAL TRIAL: NCT06554717
Title: Tesamorelin as an Adjunct to Exercise for Improving Physical Function in HIV
Acronym: TRIUMPH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Lindsay Fourman, MD, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024P001703
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: HIV-1-infection; Frailty; Impaired Physical Function; Abdominal Obesity; Aging
MeSH Terms: conditions — Frailty; Obesity, Abdominal | interventions — tesamorelin; Ghrelin; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tesamorelin Plus Exercise (Active Comparator): Tesamorelin WR 1.28 mg given subcutaneously daily plus home-based semi-supervised exercise intervention
  Interventions: Drug: Tesamorelin; Behavioral: Exercise
- Placebo Plus Exercise (Placebo Comparator): Identical placebo given subcutaneously daily plus home-based semi-supervised exercise intervention
  Interventions: Drug: Placebo; Behavioral: Exercise

INTERVENTIONS:
Drug: Tesamorelin — Tesamorelin WR 1.28 mg given subcutaneously daily
  Other Names: Egrifta, TH9507, growth hormone-releasing hormone analogue
  Arms: Tesamorelin Plus Exercise
Drug: Placebo — Identical placebo injection given subcutaneously daily
  Arms: Placebo Plus Exercise
Behavioral: Exercise — Home-based semi-supervised exercise program

SUMMARY:
People with HIV experience earlier impairments in physical function compared to people in the general population. They also exhibit an earlier presentation and more rapid development of frailty, a multisystemic syndrome of aging characterized by reduced activity, fatigue, slowness, weakness, and weight loss. While exercise can improve physical function in people with HIV, it is less effective in doing so than in the general population and is difficult to sustain in the long-term.

The goal of this clinical trial is to learn whether the medication tesamorelin will improve physical function and muscle health in adults with HIV when combined with exercise. Tesamorelin is a growth hormone-releasing hormone analogue that is FDA-approved to treat abdominal fat accumulation in people with HIV. While tesamorelin has also been shown to increase muscle mass and improve measures of muscle health, its effects on physical performance and muscle strength have not yet been evaluated.

During a 24-week intervention phase, half of participants will be randomly assigned to receive tesamorelin and half of participants will be randomly assigned to receive placebo (a look-alike substance that contains no drug). All participants also will engage in a home-based exercise intervention supervised by an exercise coach. During a subsequent 24-week extension phase, individuals will be monitored off study drug and supervised exercise, and be encouraged to continue to exercise independently.

The investigators will investigate effects of tesamorelin on physical function, muscle mass and quality, quality of life, and exercise adherence and self-efficacy. They also will evaluate whether effects of tesamorelin are maintained following treatment cessation. This study may identify an important strategy to improve how individuals aging with HIV function and feel with potential applications to other patient populations.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, 50-80 years old
2. Documented HIV infection on suppressive antiretroviral therapy for at least 1 year with HIV-1 RNA <200 copies/mL and CD4+ T cell count >200/µL 3
3. Sedentary lifestyle, defined as self-reported physical activity that breaks a sweat <3 days/week with no regular resistance exercise in the past 3 months
4. ≥1 Fried frailty criterion (weakness, slow gait speed, exhaustion, decreased physical activity, or unintentional weight loss as defined by specific thresholds)
5. Waist circumference ≥102 cm in men and ≥88 cm in women
6. Normal mammogram within 2 years (females ≤74 years old) or prostate specific antigen <4 ng/mL (males ≤70 years old) per U.S. Preventive Services Task Force (USPSTF) age-appropriate cancer screening guidelines
7. For females, postmenopausal defined as no menses for ≥12 months and anti-müllerian hormone (AMH) <20 pg/mL or history of bilateral oophorectomy at least 3 months ago
8. Provider approval to participate

Exclusion Criteria:

1. Use of tesamorelin or other growth hormone (GH)-based therapy within 6 months
2. Insulin-like growth factor 1 (IGF-1) z-score >2.0
3. HbA1c >8%
4. Active or suspected malignancy (with the exception of non-melanoma skin cancer) within 24 months
5. Supraphysiologic testosterone or corticosteroid exposure, or change in exogenous testosterone or corticosteroid dose within 3 months
6. Change in glucose-lowering medication (e.g., glucagon-like peptide-1 receptor agonists) within 3 months
7. Active or unstable coronary artery disease, chest pain suspicious for angina, or serious arrythmia
8. History of hypopituitarism, head irradiation, or other conditions known to affect the GH/IGF-1 axis
9. Known hypersensitivity to tesamorelin or mannitol
10. Acute or chronic illness judged by the investigator to represent a contraindication to study participation

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Repeated Chair Stand Time | Baseline to Week 24
  Time to complete 10 repeated chair stands

SECONDARY OUTCOMES:
Change in Standard and Modified Short Physical Performance Battery (SPPB) | Baseline to Week 24
  Objective assessment of physical function that includes measures of balance, gait, and strength
Change in 1-Repetition Maximum Leg Press | Baseline to Week 24
  Maximal weight that can be lifted by lower extremities once using correct form through full range of motion
Change in 400-Meter Walk Time | Baseline to Week 24
  Time to walk 400 meters at the fastest pace possible
Change in Appendicular Lean Tissue Mass | Baseline to Week 24
  Dual-energy x-ray absorptiometry (DXA) lean tissue mass in all four extremities
Change in Cross-Sectional Area of Trunk and Thigh Muscles | Baseline to Week 24
  Computed tomography (CT) cross-sectional area of trunk and thigh muscles
Change in Frailty Phenotype | Baseline to Week 24
  Fried Frailty Phenotype score, scored from 0 to 5 with higher indicating worse
Change in Quality of Life | Baseline to Week 24
  36-Item Short Form Health Survey (SF-36), scored from 0 to 100 with higher indicating better
Change in Exercise Self-Efficacy | Baseline to Week 24
  Exercise Self-Efficacy Scale, scored from 0 to 100 with higher indicating better
Change in Exercise Adherence | Baseline to Week 24
  FitBit (step count heart rate time), exercise log (movement type, repetitions, load, rate of perceived exertion)
Change in Tissue Density of Trunk and Thigh Muscles | Baseline to Week 24
  Computed tomography (CT) attenuation of trunk and thigh muscles
Change in Visceral Adipose Tissue Cross-Sectional Area | Baseline to Week 24
  Computed tomography (CT) cross-sectional area at L4

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay T. Fourman, MD, Principal Investigator — Massachusetts General Hospital; Kristine M. Erlandson, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado - Anschutz Medical Campus, Aurora, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts